CLINICAL TRIAL: NCT06896994
Title: Intravenous Infusion of Esketamine in Combination With Pregabalin and Duloxetine for Postherpetic Neuralgia
Brief Title: Esketamine Combined Pregabalin and Duloxetine for Postherpetic Neuralgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Xiaotangshan Hospital (Other); The First Hospital of Fangshan District,Beijing (Other); Beijing Ditan Hospital (Other); Hengshui People's Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, The Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2024-332-02-02
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Postherpetic Neuralgia
Keywords: Postherpetic Neuralgia; esketamine
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the esketamine group (Experimental): In the esketamine group, in addition to receiving the combination of pregabalin and duloxetine, patients will also undergo a single intravenous infusion of esketamine. A total of 0.5 mg/kg of esketamine will be diluted in 50 mL of normal saline. The infusion will commence with an intravenous injection of 10 mg of esketamine over 1 minute, followed by a maintenance dose of 8 mg/h. The infusion rate will be adjusted based on the patients' tolerance levels.
  Interventions: Drug: esketamine group
- the control group (Placebo Comparator): In the control group, patients will receive pregabaline combined with duloxetine. Pregabaline will be administered at a dose of 50-75 mg, twice daily during the first 3 days of treatment, and increase to 300mg daily after 3-7days, then by an additional 150mg daily every 3-7 days as tolerated, up to a maximum daily dose of 600mg. Meanwhile, duloxetine will be prescribed at an initial daily dose of 30mg, and then gradually increased to 60 mg daily after one week if patients tolerate it well.
  Interventions: Drug: control group

INTERVENTIONS:
Drug: esketamine group — In the esketamine group, in addition to receiving the combination of pregabalin and duloxetine, patients will also undergo a single intravenous infusion of esketamine.
  Other Names: pregabalin+duloxetine+esketamine
  Arms: the esketamine group
Drug: control group — receiving the combination of pregabalin and duloxetine
  Other Names: pregabalin+duloxetine
  Arms: the control group

SUMMARY:
To assess the 1-week effects and safety of esketamine in combination with pregabalin and duloxetine to relieve pain in patients with postherpetic Neuralgia(PHN).

DETAILED DESCRIPTION:
The investigators aim to investigate whether or not esketamine combined with pregabalin and duloxetine to relieve pain in patients with PHN, and seek a rapid, effective and safe treatment for refractory patients with PHN

ELIGIBILITY:
Inclusion Criteria:

1. Ages more than 18 years;
2. Pain present for more than 3 months after healing of a herpes zoster skin rash;
3. Has an average pain score of at least 4 on a Numeric Rating Scale (NRS, 0= no pain, 10= worst possible pain)；
4. Failed to respond to or tolerate the effective dose of pregabalin monotherapy.

Exclusion Criteria:

1. Obstructive sleep apnoea syndrome;
2. Those who receive interventional treatments;
3. A history of systemic immune diseases, organ transplantation, or cancers;
4. A history of severe cardiopulmonary, hepatic or renal dysfunction;
5. A history of schizophrenia, epilepsy, or myasthenia gravis, delirium;
6. Currently using monoamine oxidase inhibitors (MAOIs);
7. Having untreated angle-closure glaucoma;
8. Those suffering from increased intracranial pressure；
9. Comorbid hyperthyroidism or phaeochromocytoma;
10. Suspected or confirmed history of drug abuse;
11. Having contraindications to esketamine, pregabaline or duloxetine;
12. Communication difficulties;
13. Women who are preparing for pregnancy, in the pregnancy or lactation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
the mean of daily pain scores | during 1 week
  the mean of daily pain scores collected during week 1 of treatment measured using the Numerical Pain Rating Scale (NRS,, 0 represents no pain, and 10 represents the most severe pain.A higher score indicates more severe pain).

SECONDARY OUTCOMES:
Averaged weekly NRS score | 1 week, 2 weeks, 3 weeks, and 1 month after treatment
  Averaged weekly NRS score of each participant.Generally, 0 represents no pain, and 10 represents the most severe pain.A higher score indicates more severe pain
percentages of patients having >50% reductions in 24-hour average pain severity during the first week | during the first week
  percentages of patients having >50% reductions
the 12-item Short-Form Health Survey (SF-12) score | 1 day, 3 days, 7 days, 2 weeks, 3 weeks, and 1 month after treatment
  Quality of life (QoL) assessed by the SF-12 score (range 0-100, with higher scores indicating better health status).
the Pittsburgh Sleep Quality Index (PSQI) score | 1 day, 3 days, 7 days, 2 weeks, 3 weeks, and 1 month after treatment
  Sleep quality measured by PSQI score (range 0-21, with higher scores indicating poorer sleep quality).
the Patient Global Impression of Change scale (PGIC) | 1 day, 3 days, 7 days, 2 weeks, 3 weeks, and 1 month after treatment
  The proportion of patients with a response of "no change", "minimally improved", "much improved" or "very much improved" on PGIC.
The Hospital Anxiety and Depression Scale (HADS) | 1 day, 3 days, 7 days, 2 weeks, 3 weeks, and 1 month after treatment
  It consists of two sub-scales. Each sub-scale consists of 7 items and each item scored from 0 to 3. A higher score indicates more severe anxiety or depression. A score of 11 or above can indicate clinically significant anxiety or depression.
Averaged weekly analgesic consumption | 1 day, 3 days, 7 days, 2 weeks, 3 weeks, and 1 month after treatment
  Averaged weekly consumption per analgesic of each participant
Safety assessments | 0 day, 1 day, 3 days, 7 days, 2 weeks,3 weeks, and 1 month after treatment
  drug-related complications,such as dizziness, somnolence, gait disturbance, nausea, fatigue, diarrhea, dry mouth, mental symptom, etc

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Not yet decided